CLINICAL TRIAL: NCT04650542
Title: Open-Label, Two-Period Phase 1 Study in Healthy Subjects to Evaluate the Potential Effect of Multiple Doses of Paroxetine on the Pharmacokinetics and Safety of HBI-3000
Brief Title: Drug-Drug Interaction Study of HBI-3000 and Paroxetine in Healthy Adult Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HUYABIO International, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBI-3000-401
Record Dates: First submitted 2020-11-13; First posted 2020-12-02 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Drug-drug Interaction
MeSH Terms: interventions — sulcardine sulfate; Paroxetine

STUDY DESIGN:
Intervention Model Description: * Experimental: HBI-3000, 350 mg, 50 mL intravenous infusion (IV) over 30 minutes on Day 1 of Period 1 and approximately 15 days later on Day 1 of Period 2
  * Paroxetine: 20 mg dose twice a day on Days 1 and 2 of Period 2, and once a day on Days 3 through 7 inclusive of Period 2
Masking Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HBI-3000 alone (Period 1) followed by HBI-3000 with Paroxetine (Period 2) (Experimental): HBI-3000: 350 mg, 50 mL intravenous infusion (IV) over 30 minutes on Day 1 of Period 1 and approximately 15 days later on Day 1 of Period 2
  Paroxetine: 20 mg dose twice a day on Days 1 and 2 of Period 2, and once a day on Days 3 through 7 inclusive of Period 2
  Interventions: Drug: HBI-3000; Drug: Paroxetine

INTERVENTIONS:
Drug: HBI-3000 — small molecule, multi-ion channel blocker
  Other Names: Sulcardine sulfate
Drug: Paroxetine — serotonin uptake inhibitor, CYP2D6 inhibitor

SUMMARY:
Drug-Drug Interaction Study of HBI-3000 and Paroxetine in Healthy Adult Male and Female Subjects

DETAILED DESCRIPTION:
This is a Phase 1 study in healthy volunteers to evaluate the potential effect of multiple doses of paroxetine on the pharmacokinetics and safety of HBI-3000. Each subject serves as his/her own control: Period 1 vs. Period 2.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult males and females

* 18 - 50 years of age
* BMI 18 - 32 kg/m2
* Subject has no clinically significant abnormality on electrocardiogram (ECG)
* Subject has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least 4 months
* Subject is willing to comply with the study restrictions, including contraception requirements

Exclusion Criteria:

* Evidence of a clinically significant disease or abnormalities, including an active, current infection or clinically significant infection within 8 weeks prior to the first dose
* Severe allergic reaction, angioedema, or anaphylaxis to drugs, or food or latex allergies
* Subject has an estimated creatinine clearance of ≤ 70 mL
* Subject has evidence of a clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations
* Subject has significant ECG abnormality, history or presence of cardiac arrhythmia or conduction abnormalities, or bradycardia (< 45 bpm)
* Subject has a history of vasovagal syncope, or symptomatic orthostatic hypotension
* Subject has as a history of or current alcohol abuse and/or other drug addiction
* Subject has received an investigational drug (including investigational vaccines) within 5 half-lives of such drug prior to Study Day 1
* Subject has received CYP2D inhibitors (e.g., fluoxetine, sertraline, duloxetine, bupropion, chloroquine, cimetidine, diphenhydramine) less than 3 weeks prior to administration of the initial dose of study drug
* Subject has suicidal thinking and behavior (suicidality) or other significant psychiatric disorders based on self-disclosure during interview (Screening visit)
* Subject has a history of acute narrow-angle glaucoma
* Subject has as any condition that would make him or her, in the opinion of the Investigator or Sponsor, unsuitable for the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-02-21 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics (PK): Maximum observed plasma concentration (Cmax) | 72 hours
  To determine the plasma Cmax of a single dose of HBI 3000 administered intravenously (IV), in the absence and the presence of CYP2D6 inhibition, achieved with multiple oral doses of paroxetine, a strong CYP2D6 inhibitor, in healthy male and female subjects. Blood samples will be taken from 0 through 72 hours after the start of HBI-3000 infusion.
Plasma pharmacokinetics (PK): Area Under the Curve (AUC) from time 0 to last measurable concentration (AUC0 - tau) | 72 hours
  To determine the plasma AUC of a single dose of HBI 3000 administered intravenously (IV), in the absence and the presence of CYP2D6 inhibition, achieved with multiple oral doses of paroxetine, a strong CYP2D6 inhibitor, in healthy male and female subjects. Blood samples will be taken from 0 through 72 hours after the start of HBI-3000 infusion.
Plasma pharmacokinetics (PK): Area Under the Curve (AUC) from time 0 to infinity (AUC0 - infinity), if data permits | 72 hours
  To determine the plasma AUC of a single dose of HBI 3000 administered intravenously (IV), in the absence and the presence of CYP2D6 inhibition, achieved with multiple oral doses of paroxetine, a strong CYP2D6 inhibitor, in healthy male and female subjects. Blood samples will be taken from 0 through 72 hours after the start of HBI-3000 infusion.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Events (TEAEs), including serious TEAEs | 25 days
  To evaluate the safety and tolerability of HBI-3000 in the absence and the presence of paroxetine, as measured by Treatment-Emergent Adverse Events (TEAEs), including serious TEAEs. TEAE is defined as follows: An AE that emerges during treatment, having been absent at pretreatment (Baseline), an AE that re emerges during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or an AE that worsens in severity during treatment relative to the pretreatment state, when the AE is ongoing. TEAEs will be recorded for approximately 25 days commencing with the start of HBI-3000 infusion.
Routine hematology and coagulation | 25 days
  To evaluate the safety and tolerability of HBI-3000 in the absence and the presence of paroxetine, as measured by routine hematology and coagulation tests, at Screening and periodically during the study, including: Hematocrit (Packed cell volume); Hemoglobin; Lymphocytes; Mean cell hemoglobin Mean cell hemoglobin concentration; Mean cell volume; Basophils; Eosinophils; Monocytes; Neutrophils; Platelet count; Red blood cell count; White blood cell count; Coagulation Tests; Prothrombin time; International normalised ratio; Partial thromboplastin time
Routine serum chemistry | 25 days
  To evaluate the safety and tolerability of HBI-3000 in the absence and the presence of paroxetine, as measured by routine serum clinical chemistry tests, at Screening and periodically during the study, including: Alanine aminotransferase; Albumin; Alkaline phosphatase; Aspartate aminotransferase; Bicarbonate; Bilirubin (total); Bilirubin (direct); Calcium; Chloride; Cholesterol; Creatine kinase; Creatinine, estimated clearance; Gamma glutamyl transferase; Triglycerides; Globulin; A/G ratio; Glucose; Magnesium; Potassium; Phosphate (inorganic); Protein (total); Sodium; Urea; Uric acid
Vitals signs | 25 days
  To evaluate the safety and tolerability of HBI-3000 in the absence and the presence of paroxetine, as measured by vitals signs including heart rate and blood pressure using an automated blood pressure device, at Screening and periodically during the study.
12-lead ECG | 25 days
  To evaluate the safety and tolerability of HBI-3000 in the absence and the presence of paroxetine, as measured by 12-lead ECG. Twelve-lead ECGs will be measured at Screening and periodically during the study using standardized equipment provided by the core ECG laboratory and reviewed locally by the Investigator. QTc interval will be calculated from Fridericia's formula.
Continuous telemetry | 8 hours beginning at the start of infusion
  To evaluate the safety and tolerability of HBI-3000 in the absence and the presence of paroxetine, as measured by monitoring via a continuous cardiac telemetry monitoring system for 8 hours commencing with the start of HBI-3000 infusion
Infusion site (local) reactions | 25 days
  To evaluate the safety and tolerability of HBI-3000 in the absence and the presence of paroxetine, as measured by observing infusion site (local) reactions for the duration of the study (approximately 25 days) commencing with the start of HBI-3000 infusion
Physical examination findings | 25 days
  To evaluate the safety and tolerability of HBI-3000 in the absence and the presence of paroxetine, as measured by examination of body systems and symptom directed examination as indicated, at Screening and during the study (approximately 25 days)
Left ventricular ejection fraction (LVEF), Exploratory | At baseline and 2 hours beginning at the start of infusion
  To evaluate the safety and tolerability of HBI-3000 in the absence of paroxetine, as measured by 2D transthoracic echocardiogram to measure changes in cardiac contractility, determined at baseline and at 30 minutes and 2 hours after the start of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, Principal Investigator — Nucleus Network; Jennifer Deering, MSN, ARNP, Principal Investigator — Spaulding Clinical
Locations (2):
- Spaulding Clinical, West Bend, Wisconsin, United States
- Nucleus Network Pty Ltd., Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No